CLINICAL TRIAL: NCT04524546
Title: Sternomental Displacement and Neck Circumference as Predictors of Difficult Airway in Obese Patients During General Anesthesia: a Prospective Observational Cohort Study
Brief Title: Sternomental Displacement Test for Predicting Difficult Airway in Obese Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Assistant Professor of Anesthesia, SICU & pain management. Kasralainy Faculty of medicine, Cairo University
Other Study IDs: Ms-141-2020
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Difficult Airway Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sterno-mental displacement test — While the patient is in sitting position, (SMD neutral) will be is measured using tape as the distance between upper borders of the manubrium sterni to the mentum with the head in a neutral position. The (SMD extension) will be then measured in the same way with the head extended on the neck. The difference between SMD extension and SMD neutral will be then calculated as sternomental displacement (SMDD).

SUMMARY:
Difficulties airway significantly contribute to the morbidity and mortality associated with anesthesia. Identifying situations and patients at risk for airway management problems is the key to optimal care and has been the focus of numerous publications. Although controversial, Body Mass Index (BMI) is considered as associated with difficult intubation in both and operating theaters. A modified measurement of SMD is obtained with the head in neutral position (SMD neutral), then the difference between SMD extension and SMD neutral was calculated and it was referred to as sternomental displacement (SMDD). SMDD was proved to be a good objective predictor for difficult laryngoscopy in adult patients, and its predictive ability was increased when combined with other tests as neck circumference (NC). To the best of our knowledge, the validity of the SMDD test was not previously assessed in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, aged between 18-60 years old, ASA physical status II & III with BMI > 30 Kg/m2 undergoing elective surgical procedures under general anesthesia using endotracheal intubation by conventional laryngoscopy.

Exclusion Criteria:

* neuromuscular disorders, craniofacial abnormalities, abnormal dentition, lesions or scares in head and neck limiting the neck mobility, uncooperative, who needed awake intubation and patients who underwent emergency operations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients of either sex, aged between 18-60 years old, ASA physical status II & III with BMI > 30 Kg/m2
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
A a cut-off value, sensitivity (Sn), specificity (Sp), positive predictive values (PPV), negative predictive values (NPV) of sternomental displacement in predicting difficult laryngoscopy in obese patient undergoing GA. | before induction of general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia department - Faculty of medicine- Cairo University, Cairo, Egypt